CLINICAL TRIAL: NCT05943314
Title: Safety and Efficacy of Anti-CLL1 /+CD33 CAR T Cells in Refractory/Recurrent Acute Myeloid Leukemia: a Single-arm, Non-blind Clinical Study
Brief Title: Clinical Study on Safety and Efficacy of Anti-CLL1 /+CD33 CAR T Cells in the Treatment of Acute Myeloid Leukemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical trial was terminated due to a change in sponsor strategy.
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-21-001
Record Dates: First submitted 2023-06-09; First posted 2023-07-13 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; CLL1; CD33
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLL1/+CD33 CAR-T (Experimental): The target dose range for subjects was set to be 1.00~2.50x10^6/kg CAR-positive T cells.
  Interventions: Biological: CLL1/+CD33 CAR-T

INTERVENTIONS:
Biological: CLL1/+CD33 CAR-T — CLL1/+CD33 CAR T is a type of CAR T cell therapy for patients with treating/relapsed acute myeloid leukemia.

SUMMARY:
This is a single-center, single-arm, open, intravenous drug administration of the safety and efficacy of clinical study.

DETAILED DESCRIPTION:
The primary objective of the clinical trial was to evaluate the safety and efficacy of single dose infusion of anti-CLL1 /+CD33 CAR T cells in patients with refractory/recurrent acute myeloid leukemia. A total of about 5 patients with refractory/recurrent acute myeloid leukemia were enrolled in this study, and the target dose range was 1.00~2.50x10^6/kgCAR-positive T cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her legal guardian volunteers for the trial and signs an informed consent form;
2. Age range 1-18 years;
3. Acute myeloid leukemia (AML) with CLL1 and CD33 markers (including secondary patients) was diagnosed by pathology, histology and flow cytometry, or complete hematologic remission could not be achieved after 1 course of chemotherapy for hematologic relapse after drug withdrawal ;
4. The main organ functions of the patients were good: (1) liver function: ALT/AST < 3 times the upper limit of normal (ULN) and bilirubin ≤34.2 μmol/l; (2) renal function: creatinine < 220 μmol/l; (3) lung function: oxygen saturation ≥95% ; (4) cardiac function: left ventricular ejection fraction (LVEF)≥40% ;
5. The blood flow of peripheral superficial vein was unobstructed, which could meet the demands of intravenous drip and mononuclear cell collection;
6. ECOG score was 0-2.

Exclusion Criteria:

1. The patients had uncontrollable infectious diseases within 4 weeks before the enrollment;
2. Active hepatitis B/C virus;
3. HIV infection, treponema syphilis positive patients;
4. Pathological diagnosis of primary tumors other than acute myeloid leukemia;
5. Suffering from serious autoimmune diseases or immunodeficiency diseases;
6. The patient is allergic to antibodies or cytokines and other macromolecular biological drugs;
7. Pregnant or lactating women;
8. Patients who were considered ineligible for study for other reasons.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Changes in cytokine level after CLL1/+CD33 CAR-T infusion | CAR T cell infusion before and 12 months after infusion
  Calculate the change of cytokine level in peripheral blood by flow cytometry after CAR-T infusion.
The change characteristics of chimeric antigen receptor(CAR)-T cell number in patients after infusion. | CAR T cell infusion before and 12 months after infusion
  Track CAR-T cells expansion in patients after infusion by flow cytometry
The change characteristics of chimeric antigen receptor(CAR)-T cell copy number in patients after infusion. | CAR T cell infusion before and 12 months after infusion
  Track CAR-T cells expansion in patients after infusion by Real-time Quantitative Polymerase Chain Reaction（qPCR）

SECONDARY OUTCOMES:
Event-free survival | Up to 12 months after CLL1/+CD33 CAR-T infusion
  Counting from the beginning of cell transfusion until treatment failure, recurrence, or death (various causes). Subjects without any of these events were counted up to the last follow-up examination date. For patients without CR or CRi, EFS is calculated from the beginning of cell transfusion until disease progression or death. Based on the initial event.
Overall survival | Up to 12 months after CLL1/+CD33 CAR-T infusion
  Death from any cause from the beginning of cell transfusion
Duration of Overall Response | Up to 12 months after CLL1/+CD33 CAR-T infusion
  The time from the start of cell infusion when CR or PR is first achieved to disease progression.
MRD negative rate | Up to 12 months after CLL1/+CD33 CAR-T infusion
  The rate of MRD negative subjects was determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, doctor, Principal Investigator — Children's Hospital of Fujian Province
Locations (1):
- Fujian Provincial Children's Hospital, Fuzhou, Fujian, China